Title: Adherence to Guidelines VAccination in Type 1 Dlabetes Mellitus Patients (AVADI-1).

NCT03478254 Unique Protocol ID: C-127.

Date: July 15th 2017

## **Study procotol:**

# **Design:**

This was a cross-sectional analysis of data extracted from the electronic medical record (EMR) system at Ciudad Real Health Public Area (Castilla-La Mancha Health Public System, Spain).

#### **Ethics:**

The protocol was approved by the reference Castilla-La Man-cha Public Health Institute Ethic Committee.

All participants provided written informed consent.

The protocol was publicly registered through Clinical Trials (NCT03478254).

#### Dates:

The study was conducted from 1 December 2017 to 1December 2018.

## **Subjects:**

All adult (≥18 years of age) patients diagnosed of T1DM from our electronic database were eligible for chart review.

## **Endpoints:**

Primary efficacy outcome was to describe influenza, pneumococcal and HBV vaccination status.

Secondary efficacy outcomes were to identify predictor of adherence to vaccination program and to analyse absence of vaccination impact (sick leaves and hospitalizations). Data collected through chart review from EMR.